CLINICAL TRIAL: NCT00716105
Title: Effect of the Level of Dietary Protein on Infant Growth and Body Composition in the First Year of Life
Brief Title: Effect of the Level of Dietary Protein on Infant Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 06.29.INF
Record Dates: First submitted 2008-07-11; First posted 2008-07-16 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2014-10

CONDITIONS: Infant Nutrition
Keywords: Infant formula; Protein metabolism
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Standard Infant Formula
  Interventions: Other: Standard infant formula
- Test Product (Experimental): Infant formula with different level of proteins
  Interventions: Other: Infant formula with different level of proteins
- Breast Milk (No Intervention): Breastfeeding reference group

INTERVENTIONS:
Other: Standard infant formula — From 3 to 12 months of age. As per standard requirement
  Arms: Control
Other: Infant formula with different level of proteins — From 3 to 12 months of age. As per standard requirement
  Arms: Test Product

SUMMARY:
The purpose of this study is to determine whether infants fed a formula with protein levels different than a standard infant formula have similar growth and development.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at least 37 weeks
* Singleton birth
* Birth weight between 2500g and 4500g
* Weight at enrolment is at or above the 5th percentile (CDC)
* Infant has been exclusively formula fed for at least the last 14 days
* Having obtained informed consent of legal representative

Exclusion Criteria:

* Congenital illness or malformation that affects infant feeding and/or growth
* Significant pre-natal and/or post-natal disease
* Suspected or confirmed allergy to cow milk protein
* In the investigators assessment, infant's family cannot be expected to comply with treatment (feeding regimen)
* Currently participating in another clinical trial

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 405 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Mean weight gain | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ekhard E Ziegler, MD, Principal Investigator — The Samuel J. Fomon Infant Nutrition Unit Dept of Pediatrics, University of Iowa
Locations (2):
- United States (2):
  - The Samuel J. Fomon Infant Nutrition Unit Dept of Pediatrics, University of Iowa, Iowa City, Iowa
  - Department of Pediatrics University of Oklahoma Health Sciences, Oklahoma City, Oklahoma

REFERENCES:
- [Derived] Ziegler EE, Fields DA, Chernausek SD, Steenhout P, Grathwohl D, Jeter JM, Nelson SE, Haschke F. Adequacy of Infant Formula With Protein Content of 1.6 g/100 kcal for Infants Between 3 and 12 Months. J Pediatr Gastroenterol Nutr. 2015 Nov;61(5):596-603. doi: 10.1097/MPG.0000000000000881. PMID 26154030